CLINICAL TRIAL: NCT01039701
Title: Safety, Tolerability and Pharmacokinetics of 3 Dose Regimens of AZD1446 vs. Placebo as an Add-on Treatment to Donepezil: A Multi-centre, Double-blind, Randomised, Placebo Controlled, Parallel Group Phase IIa Study in Patients With Mild to Moderate Alzheimer's Disease During 4 Weeks of Treatment
Brief Title: 4 Week, Safety and Tolerability Study in Patients With Mild to Moderate Alzheimer's Disease
Acronym: ROBIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D1950C00006
Record Dates: First submitted 2009-12-20; First posted 2009-12-25 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Mild to Moderate Alzheimer's Disease
Keywords: safety; tolerability; mild to moderate Alzheimer's disease; To determine the safety and tolerability of AZD1446 vs Placebo given as an add-on treatment to Donepezil in patients with mild to moderate Alzheimer's disease
MeSH Terms: interventions — 3-(5-chloro-2-furoyl)-3,7-diazabicyclo(3.3.0)octane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): AZD1446 60mg once daily + donepezil 10mg
  Interventions: Drug: AZD1446
- 2 (Experimental): AZD1446 60mg three times daily + donepezil 10mg
  Interventions: Drug: AZD1446
- 3 (Experimental): AZD1446 30mg three times daily + donepezil 10mg
  Interventions: Drug: AZD1446
- 4 (Placebo Comparator): placebo + donepezil 10mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1446 — capsules, oral, 3 times daily
  Arms: 1; 2; 3
Drug: Placebo — capsules, oral, 3 times daily, 4 weeks
  Arms: 4

SUMMARY:
The primary purpose of the study is to determine the safety and tolerability of AZD1446 vs Placebo given as an add-on treatment to Donepezil for 4 weeks in patients with mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* history of progressive worsening of memory and other cognitive functions for at least 12 months
* treatment with stable dose of donepezil (10 mg) for at least 3 months
* the patient should have an appropriate caregiver, who is required for all study visits

Exclusion Criteria:

* history of allergy/hypersensitivity reactions
* significant neurological disease or dementia other than Alzheimer's disease
* myocardial infarction or acute coronary syndrome within the last year

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2009-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Nature and incidence of adverse events | From the enrollment visit until the last study follow-up visit. The measure will be taken at each scheduled study visit and in between visits , if any adverse events occur.

SECONDARY OUTCOMES:
To evaluate any effects PK of AZD1446 as an add-on treatment to donepezil on the PK of donepezil | Twice during the study: at Visit 2 and Visit 10.
To characterize the PK of AZD1446 as an add-on treatment to donepezil in AD patients | Twice during the study: at Visit 8 and Visit 10.
To explore the effects of 3 dose regimens of AZD1446 compared to placebo as an add-on treatment to donepezil on changes in global functioning using ADCS-CGIC | Baseline assessment at Visit 2 and a follow-up assessment at Visit 10

CONTACTS AND LOCATIONS:
Locations (12):
- Czechia (3):
  - Research Site, Litoměřice
  - Research Site, Prague
  - Research Site, Praha 10 - Strasnice
- Hungary (6):
  - Research Site, Debrecen
  - Research Site, Esztergom
  - Research Site, Miskolc
  - Research Site, Nagykálló
  - Research Site, Nyíregyháza
  - Research Site, Szeged
- Slovakia (3):
  - Research Site, Bratislava
  - Research Site, Rožňava
  - Research Site, Zlaté Moravce